CLINICAL TRIAL: NCT00678158
Title: Phase I Dose Escalation Study Using High-Dose Single Fraction Image-Guided Radiotherapy for Metastatic Lesions to Soft Tissue Masses, Lymph Node, or Bone
Brief Title: Study Using High-Dose Single Fraction Image-Guided Radiotherapy for Metastatic Lesions to Soft Tissue Masses, Lymph Node, or Bone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-101
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Disease
Keywords: High Does Single Fraction IGRT; Bone; Lymph Nodes; Soft Tissue
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiotherapy, Intensity-Modulated

ARMS (3):
- 1 (Experimental): Patients with metastatic disease to soft tissue.
  Interventions: Radiation: intensity modulated radiation therapy
- 2 (Experimental): Patients with metastatic disease to lymph nodes.
  Interventions: Radiation: intensity modulated radiation therapy
- 3 (Experimental): Patients with metastatic disease to the bone.
  Interventions: Radiation: intensity modulated radiation therapy

INTERVENTIONS:
Radiation: intensity modulated radiation therapy — Patients will be accrued at each dose level beginning at 22 Gy with increments of 2 Gy up to 28 Gy. Patients with a soft tissue mass, lymph nodes or focal bone metastases with lesions large enough to be imaged on CT scan will be accrued. Starting at 24 Gy, patients will be stratified in to 3 treatment categories: lesions involving bone, bowel, or spinal cord. Patients will be enrolled in each treatment category until 10 patients in that cohort reach an evaluable timepoint of 3 months post-RT. The maximum accrual is 20 for 22 Gy, and 90 (30 per treatment category) for each subsequent dose level (24-28 Gy). Some of these patients have participated in the optional FLT-PET scan portion of the study. Some of these patients have under gone an optional MRI scan which take place within one hour of the radiation treatment .

SUMMARY:
The purpose of this research study is to find out what IG-IMRT radiation dose works best for treatment of disease in bone or soft tissues. This protocol will study what dose level may work most effectively. The first part of study will treat 10 patients with 22 Gray. Gray (Gy) is the unit that is used to describe the dose of radiation that is being given to a person with cancer. After we confirm that 22 Gy is a safe and sufficient amount of radiation, we will then treat another group of patients with 24 Gy and so on until we reach 28 Gy. Each dose level starting with 24 Gy will enroll at least 20 patients per treatment site (bone, bowel and/or spine). Patients will be enrolled in each treatment category until 20 patients in each strata reach an evaluable time point of 3 months post-RT. When we understand what dose works best and has the least amount of bad effects, the study will then look to see how well the patients do after the radiation therapy. This study is trying to see how your doctor can best treat the cancer that has spread to the other parts of your body.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven cancer verified at MSKCC
* Imaging evidence of lymph node metastases, bone metastases or soft tissue disease
* Age > or = to 18 years
* KPS > or = to 80
* Epidural disease is acceptable as long as the dose to the spinal cord ≤ 14 Gy
* Able to tolerate immobilization cradle positioning

Exclusion Criteria:

* Target lesion not visible on conventional CT scan
* Unable to be administered intravenous CT contrast safely
* Prior radiation to the planned target region. A second metastatic lesion would not be eligible if the area received or will receive any dose (5% or greater isodose line)from a prior or planned single fraction treatment
* Patients receiving concurrent chemotherapy (within 1 week of RT)
* Normal tissue directly overlying target precluding ability to limit the bowel, bladder, rectum or other tissue to 15-16 Gy dose constraints
* Weight-bearing bones with significant cortical destruction from tumor. In these cases, patients will be referred for orthopedic consultation for rod stabilization procedures.
* Subjects with more than 4 metastases to bone
* Any metastatic lesion larger than 8 cm in its greatest diameter

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of single dose image-guided intensity modulated radiotherapy (IGIMRT)for metastatic disease to soft tissue, lymph nodes or bones. | conclusion of the study

SECONDARY OUTCOMES:
To establish the maximal safe single fraction dose for osseous and soft tissue metastatic lesions using IG-IMRT in a Phase I dose escalation study. | conclusion of the study
To obtain information on the effect of high-dose external beam irradiation on the biodistribution and pharmacokinetics of FLT. | 2 years
To obtain preliminary information on the changes in tumor perfusion resulting from high-dose, single fraction IGRT for patients treated with approach to focal metastases using dynamic contrast-enhanced (DCE)-MRI. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zelefsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org